CLINICAL TRIAL: NCT03324529
Title: Autonomic Modulation in Takotsubo Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00868
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants in the NYU takotsubo registry (Experimental): 10 patients with a confirmed history of takotsubo syndrome
  10 age- and sex-matched healthy controls with no significant history of cardiac or neurological illness
  Interventions: Device: Tako Breath

INTERVENTIONS:
Device: Tako Breath — Device guided breathing. A medical device with a computerized control unit, a breathing sensor and a set of earphones with audio-prompts to guide breathing at a slow rate (<10 breaths/min) with prolonged exhalation.
  Other Names: RESPeRATE

SUMMARY:
This is a minimal risk case-controlled single arm intervention study, including 10 patients with a prior history of takotsubo and 10-age and sex matched healthy controls. Subjects will undergo in laboratory testing to measure autonomic function. They will then undergo a 15-week program of device-guided breathing with remote measures of autonomic function obtained at home. Analysis will determine the reproducibility of home autonomic measures and the provide preliminary data to determine the efficacy of device-guided breathing on autonomic measures and quality of life in patients with takotsubo.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed history of takotsubo syndrome
* Healthy person with no significant past history of cardiovascular or neurological disease such as heart failure or heart attack; people with cardiovascular risk factors such as hypertension will be permitted to participate

Exclusion Criteria:

* Pacemaker or defibrillator implanted
* Evidence of autonomic neuropathy, alcohol or drug abuse or exposure to neurotoxins (chemotherapy).
* Diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | 10 Weeks
  Remote heart rate monitoring with an adhesive chest telemetry patch and biosensor wrist watch

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No